CLINICAL TRIAL: NCT03248310
Title: A Prospective Study Comparing Quality of Life in Patients With Lymphedema Who Undergo Surgical Treatment Versus Non-Surgical Management
Brief Title: A Study Comparing Quality of Life in Patients With Lymphedema Who Undergo Surgical Treatment Versus Non-Surgical Management
Status: Recruiting | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 17-377
Record Dates: First submitted 2017-08-10; First posted 2017-08-14 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Lymphedema
Keywords: Quality of Life (QoL); 17-377
MeSH Terms: conditions — Lymphedema

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- vascularized lymph node transfer (VLNT): This is an observational study to assess QOL in patients who have elected to undergo or considered undergoing VLNT. There is no therapeutic intervention involved during the follow-up study period.
  Interventions: Behavioral: Quality of Life Assessments
- non-surgical treatment: This is an observational study to assess QOL in patients who have elected to undergo or considered undergoing VLNT. There is no therapeutic intervention involved during the follow-up study period.
  Interventions: Behavioral: Quality of Life Assessments

INTERVENTIONS:
Behavioral: Quality of Life Assessments — Upper Limb Lymphedema (ULL-27), Lymphedema Life Impact Scale, version 2 (LLISv2), LYMQOL-Leg.

SUMMARY:
This study is being done to see the long-term results for patients who choose to have surgery for lymphedema (with the vascularized lymph node transfer), compared to patients who choose not to have surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-80 years
* Primary and secondary lymphedema of the upper or lower extremity
* International Society of Lymphology (ISL) Stage 1, 2, or 3 lymphedema
* Proficiency in English language

Exclusion Criteria:

* Patients with clotting disorders, venous insufficiency, end-stage lymphedema unless they are on the non-surgical arm.
* Additionally, if the patient refuses to complete questionnaires, the patient will be excluded from the study and replaced at the discretion of the principal or co-principal investigator.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients who present for consultation of their lymphedema and who meet eligibility criteria will be offered the option of enrolling in this study at the time of their initial consultation.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2017-08-09 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Quality of Life | up to 40 months
  Questionnaire to assess quality of life changes

CONTACTS AND LOCATIONS:
Overall Officials: Babak Mahrara, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (3):
- United States (3):
  - Memorial Sloan Kettering Westchester (Limited Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau (Limited Protocol Activites), Rockville Centre, New York

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm